CLINICAL TRIAL: NCT01524822
Title: Experienced Breacher Study: Evaluation of the Effects From Chronic Exposure to Low-Level Blast
Brief Title: The Effects of Chronic Exposure to Low-Level Blasts
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120065; 12-N-0065
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2023-03-14

CONDITIONS: Tramatic Brain Injury
Keywords: Military; Traumatic Brain Injury; Cognitive Testing; Neuroimaging; Natural History; Brain Function
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Artillery personnel: exposure to a significant number of concussive evolutions, specifically, exposure to 400 or more within a career, will be considered experienced by the investigators.
- Breachers: exposure to a significant number of breaching blasts, specifically, exposure to 400 breaching blasts or more within a career, will be considered experienced by the investigators
- Companions: The criterion is met by a person who has both some historical knowledge of the participant and routine interactions outside a work environment.
- Unexposed: People not exposed to repeated blasts

SUMMARY:
Background:

- Repeated exposure to explosions may lead to changes in the way that people think or feel. Breachers (people trained to use explosives to get into buildings) are exposed to repeated blasts as part of their job. Researchers want to study how they might be affected by blast exposure. Breachers will be compared with other groups who have different levels of exposure to repeated blasts. Information will also be obtained from spouses or close companions.

Objectives:

- To study the effects of repeated exposure to low-level blasts on thinking, memory, behavior, and brain function.

Eligibility:

* Experienced military and civilian breachers, experienced active duty artillery operators, and active duty military without frequent blast exposure, 18 and 60 years of age.
* Spouses or close companions of these individuals.

Design:

* Participants will be screened with a physical exam and medical history. Blood samples will be collected and a urine pregnancy test will be required of participants (not companions) before MRI scanning.
* Participants will spend up to 5-days as a NIH clinic outpatient, with about 6 hours of tests each day. Tests will include the following:
* Medical and professional history, with questions about exposures to blasts
* Tests of thinking, memory, and concentration
* Balance tests
* Hearing tests
* Imaging studies, such as magnetic resonance imaging, to look at the brain
* Overnight sleep study to monitor brain waves
* Blood samples
* Participants will return 1 year later for a 3-day followup visit. Some of the tests from before will be repeated. A spouse or close companion (if available) will be asked to complete questionnaires or have a telephone interview....

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the cognitive and neurophysiological effects of chronic exposure to repeated low-level blast overpressure. Previous studies show converging evidence for a neurophysiological effect from cumulative exposure to blast, which is consistent with subjective reports of cognitive impairment by individuals trained to use explosives to gain entry to structures (breachers). This study will expand on these findings by examining a larger cohort of experienced breachers and artillery personnel who may be incurring a cumulative effect of low-level blast exposure over the course of several years. We will evaluate up to 20 participants from each of three groups: breachers, artillery personnel, and unexposed individuals. Additionally, we will ask each of the above to bring a close companion for a set of questionnaires and an interview to capture changes in functioning that participants may not be able to self-assess. Participants will travel to the NIH for evaluation of cognitive and neurophysiological measures. The procedures include neuropsychological testing, blood analysis for biomarkers, vestibular and auditory testing, and neuroimaging studies using diffusion tensor imaging, susceptibility weighted imaging, perfusion imaging, functional magnetic resonance imaging, and, where there is evidence of a sleep disorder, polysomnography. This study will be conducted in collaboration with the Naval Medical Research Center (NMRC) and the Walter Reed Army Institute of Research (WRAIR) under a Research Collaborative Agreement. The complementary DoD protocol will be reviewed by the DoD IRB and includes this NIH protocol. The complementary DoD protocol includes data collection at field settings, activity NIH is not engaged in and not described in this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

EXPERIMENTAL GROUP: BREACHERS

* Active duty and veterans who have left active duty within the previous five years or civilian law enforcement personnel
* Ages 18 60 (age range for an active duty military population)
* At least 4 years of experience in the breaching profession and actively involved in breacher training and/or operations (minimum of annual exposure). An alternate criterion to years of breacher experience is exposure to a significant number of breaching blasts, specifically, exposure to 400 breaching blasts or more within a career, will be considered experienced by the investigators.

EXPERIMENTAL GROUP 2: ARTILLERY

* Active duty and veterans who have left active duty within the previous five years
* Matched to the breacher group in terms of age, gender, and operational experience. Operational experience is defined as years of experience actively involved in artillery operations and/or number of artillery evolutions.
* At least 4 years experience with exposure to concussive environments not related to blast (minimum of annual exposure). An alternate criterion to years of experience is exposure to a significant number of concussive evolutions, specifically, exposure to 400 or more within a career, will be considered experienced by the investigators.

CONTROL GROUP: UNEXPOSED

* Active duty and veterans who have left active duty within the previous five years
* Matched to the experimental group (breachers) in terms of age, gender, and operational experience. Operational experience is defined as years of experience actively involved in military or law enforcement operations with the condition that operations include direct mission engagement roles rather than support roles. Military deployment or law enforcement patrol are examples of direct mission engagement roles and shore logistics or office based call center are examples of support roles.

COMPANION GROUP

* Spouse, close family member, or other living partner of an experimental or control group participant. The criterion is met by a person who has both some historical knowledge of the participant and routine interactions outside a work environment.
* Over 18 years of age
* Knowledge of the experimental or control group participant s daily functioning
* Companions who are unable to travel to NIH may participate remotely ( off-site companion )

EXCLUSION CRITERIA:

BREACHERS

* History of moderate or more severe brain injury with loss of consciousness greater than 5 minutes
* Current diagnosis of other CNS disorder (mild to severe)
* Any cardiac, respiratory, or other medical condition that may affect cerebral metabolism
* MRI contraindications

  * Metal in the body which would make having an MRI scan unsafe, such as pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent eye liner or small metal fragments in the eye
  * Claustrophobia
  * Inability to lie supine for up to 2 hours in the MRI scanner

ARTILLERY & UNEXPOSED

-Parallel to exclusion criteria for the breacher group, with the addition of exposure to breaching blast (greater than 40 individual blasts) for the Artillery Group and exposure to any blast (greater than 40 individual blasts) for the Unexposed Group.

COMPANION GROUP

-None

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 120 total: 20 breachers, 20 artillery, 20 unexposed controls, and 60 companions
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2012-07-30 (Actual)

PRIMARY OUTCOMES:
computer-based standardized testing, specifically the ANAM battery and the Simple Reaction Time (SRT) subtest within that battery | 10 years
  The primary objective for this study is based on anecdotal report of blast-related symptomology and previous and ongoing studies with the breacher community, suggesting a relation between post-concussive symptomology and chronic exposure to low yield blast. Measures employed in this protocol are based on measures used in other protocols in this line of research, measures used inmilitary clinical practice for concussion, and measures outlined in literature as sensitive to brain injury. These include neuroimaging procedures (fMRI, DTI, SWI, and Gadolinium contrast), neurocognitive testing, and vestibular testing.

SECONDARY OUTCOMES:
blood draw and analysis for biomarkers of brain injury and tests of peripheral auditory functioning and polysomnography to address potential confounds. | 10 years
  The secondary objectives for this study are intended to be complementary to the primary research questions and are considered important supporting data. These include blood analysis for biomarkers of brain injury, tests of peripheral auditory functioning, and polysomnography.

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Basford JR, Chou LS, Kaufman KR, Brey RH, Walker A, Malec JF, Moessner AM, Brown AW. An assessment of gait and balance deficits after traumatic brain injury. Arch Phys Med Rehabil. 2003 Mar;84(3):343-9. doi: 10.1053/apmr.2003.50034. PMID 12638101
- [Background] Bonnet MH, Arand DL. EEG arousal norms by age. J Clin Sleep Med. 2007 Apr 15;3(3):271-4. PMID 17561594
- [Background] El-Kashlan HK, Shepard NT, Asher AM, Smith-Wheelock M, Telian SA. Evaluation of clinical measures of equilibrium. Laryngoscope. 1998 Mar;108(3):311-9. doi: 10.1097/00005537-199803000-00002. PMID 9504600
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-N-0065.html